CLINICAL TRIAL: NCT02829190
Title: Feasibility Study of Phase-contrast MRI for Flow in the External Carotid Branches Arteries in Normal and Pathological Cases
Brief Title: Feasibility Study of Phase-contrast MRI for Flow in the External Carotid Branches Arteries
Acronym: IRM-de-FLUX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2013_843_0006; 2013-A00319-36 (Other: ID-RCB)
Record Dates: First submitted 2014-12-01; First posted 2016-07-12 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Carotid Artery, External
Keywords: External carotid artery; Facial artery; Lingual artery; Superior thyroid artery; Internal maxillary artery; Phase-contrast MRI; Rate of flow; Superficial temporal artery
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy volunteers (Experimental): Magnetic Resonance Imaging (MRI)
  Interventions: Device: Magnetic Resonance Imaging (MRI),
- Patients treated by radiotherapy (Experimental): Magnetic Resonance Imaging (MRI)
  Interventions: Device: Magnetic Resonance Imaging (MRI),
- Patients treated by embolization (Experimental): Magnetic Resonance Imaging (MRI)
  Interventions: Device: Magnetic Resonance Imaging (MRI),
- Patient operated on with free flap (Experimental): Magnetic Resonance Imaging (MRI)
  Interventions: Device: Magnetic Resonance Imaging (MRI),

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI), — Magnetic Resonance Imaging (MRI) of flow using phase contrast (PC) methods

SUMMARY:
The phase-contrast MRI offers the advantage to combine precisely vascular flow measurements data with morphological images.

Even if the anatomy of the external carotid artery is well known, data obtained through Phase contrast MRI could permit to progress in several fields of cranio-maxillofacial surgery as for example arteriovenous malformations,radionecrosis, head and neck micro-reconstructive surgery.

The aim of this study is to establish and develop Phase-contrast MRI sequences for vascular flow characterization branches of the external carotid artery in healthy patients and in pathological cases.

ELIGIBILITY:
Inclusion Criteria:

* group 1 : healthy volunteer
* group 2 : X-Ray treatment antecedent (at least 50 grays and older than one year)
* group 3 : antecedent of embolization of branches of external carotid artery
* group 4 : antecedent of muscular free flap surgery (older than one month)
* free and informed consent

Exclusion Criteria:

* group 1 : facial pathology, antecedent of facial injury, antecedent of X-Ray treatment in head and neck localisation, antecedent of head and neck cancer
* group 2 : antecedent of surgery for head and neck cancer or for vascular disease
* group 3 : antecedent of surgery for head and neck cancer or for vascular disease ; antecedent of X-Ray treatment.
* group 4 : antecedent of surgery for head and neck cancer or for vascular disease ; antecedent of X-Ray treatment or embolization
* patient with guardianship or trusteeship
* MRI cons-indications
* pregnancy and lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
measurability of flow 1 | 1 hour
  flow data in the branches of external carotid artery in every 4 groups, characterized by measuring the maximum speed
measurability of flow 2 | 1 hour
  flow data in the branches of external carotid artery in every 4 groups, characterized by measuring the minimum speed
measurability of flow 3 | 1 hour
  flow data in the branches of external carotid artery in every 4 groups, characterized by measuring the average speed
measurability of flow 4 | 1 hour
  flow data in the branches of external carotid artery in every 4 groups, characterized by measuring the maximum flow rates
measurability of flow 5 | 1 hour
  flow data in the branches of external carotid artery in every 4 groups, characterized by measuring the minimal flow rates
measurability of flow 6 | 1 hour
  flow data in the branches of external carotid artery in every 4 groups, characterized by measuring the medium flow rates

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DEVAUCHELLE, MD, phD, Principal Investigator — Amiens University Hospital
Locations (1):
- Departement of Maxillo-Facial Surgery, Amiens University Hospital, Amiens, Picardie, France

REFERENCES:
- [Background] Baledent O, Fin L, Khuoy L, Ambarki K, Gauvin AC, Gondry-Jouet C, Meyer ME. Brain hydrodynamics study by phase-contrast magnetic resonance imaging and transcranial color doppler. J Magn Reson Imaging. 2006 Nov;24(5):995-1004. doi: 10.1002/jmri.20722. PMID 17024656
- [Background] Cadenat H, Barthelemy R, Combelles R, Fabie M, Maneaud M. [Importance of mandibular vascularization in maxillofacial surgery]. Rev Stomatol Chir Maxillofac. 1972 Jan-Feb;73(1):60-5. No abstract available. French. PMID 4504634
- [Background] Castelli WA, Nasjleti CE, Diaz-Perez R. Interruption of the arterial inferior alveolar flow and its effects on mandibular collateral circulation and dental tissues. J Dent Res. 1975 Jul-Aug;54(4):708-15. doi: 10.1177/00220345750540040301. PMID 808564
- [Background] Combelles R, Manelfe C, Hugot B, Pasturel J, Barthelemy R, Fabie M, Cadenat H. [Selective catherization of the external carotid in stomatology]. Rev Odontostomatol Midi Fr. 1974;32(1):19-37. No abstract available. French. PMID 4438882
- [Background] Dakpé, S., 2007. Allotransplantation faciale composite: reflexion à propos de l'intégration de trois greffons expérimentaux.Université Paris XI.
- [Background] Decorato I, Kharboutly Z, Vassallo T, Penrose J, Legallais C, Salsac AV. Numerical simulation of the fluid structure interactions in a compliant patient-specific arteriovenous fistula. Int J Numer Method Biomed Eng. 2014 Feb;30(2):143-59. doi: 10.1002/cnm.2595. Epub 2013 Nov 5. PMID 24493402
- [Background] d'Hauthuille C, Testelin S, Moure C, Gbaguidi C, Devauchelle B. [Mandibular osteoradionecrosis. Part II: efficiency of revascularization surgery]. Rev Stomatol Chir Maxillofac. 2008 Nov;109(5):296-300. doi: 10.1016/j.stomax.2007.12.009. Epub 2008 Jun 4. French. PMID 18534648
- [Background] Frydrychowicz A, Francois CJ, Turski PA. Four-dimensional phase contrast magnetic resonance angiography: potential clinical applications. Eur J Radiol. 2011 Oct;80(1):24-35. doi: 10.1016/j.ejrad.2011.01.094. Epub 2011 Feb 17. PMID 21333479
- [Background] Gauvrit J, Trystram D, Oppenheim C, Leclerc X. [Advanced vascular imaging techniques of supra-aortic, encephalic and medullary vessels]. J Radiol. 2007 Mar;88(3 Pt 2):472-82. doi: 10.1016/s0221-0363(07)89847-7. French. PMID 17457258
- [Background] Herment A, Lefort M, Kachenoura N, De Cesare A, Taviani V, Graves MJ, Pellot-Barakat C, Frouin F, Mousseaux E. Automated estimation of aortic strain from steady-state free-precession and phase contrast MR images. Magn Reson Med. 2011 Apr;65(4):986-93. doi: 10.1002/mrm.22678. Epub 2010 Nov 3. PMID 21413062
- [Background] Houseman ND, Taylor GI, Pan WR. The angiosomes of the head and neck: anatomic study and clinical applications. Plast Reconstr Surg. 2000 Jun;105(7):2287-313. doi: 10.1097/00006534-200006000-00001. PMID 10845282
- [Background] Maurits NM, Loots GE, Veldman AE. The influence of vessel wall elasticity and peripheral resistance on the carotid artery flow wave form: a CFD model compared to in vivo ultrasound measurements. J Biomech. 2007;40(2):427-36. doi: 10.1016/j.jbiomech.2005.12.008. Epub 2006 Feb 7. PMID 16464454
- [Background] Morita S, Suzuki K, Masukawa A, Kojima S, Hirata M, Ueno E. Identification of efferent flow in the superior vena cava and azygos vein confluence using cine phase-contrast MRI: speculation of the role of the azygos arch valves. Magn Reson Imaging. 2010 Nov;28(9):1306-10. doi: 10.1016/j.mri.2010.06.005. Epub 2010 Aug 4. PMID 20685054
- [Background] Mouton Paradot G, Baledent O, Sallioux G, Lehmann P, Gondry-Jouet C, Le Gars D. [Contribution of phase-contrast MRI to the management of patients with normal pressure hydrocephalus: Can it predict response to shunting?]. Neurochirurgie. 2010 Feb;56(1):50-4. doi: 10.1016/j.neuchi.2009.12.007. Epub 2010 Jan 25. French. PMID 20097391
- [Background] Nayler GL, Firmin DN, Longmore DB. Blood flow imaging by cine magnetic resonance. J Comput Assist Tomogr. 1986 Sep-Oct;10(5):715-22. doi: 10.1097/00004728-198609000-00001. PMID 3528245
- [Background] Pomahac B, Lengele B, Ridgway EB, Matros E, Andrews BT, Cooper JS, Kutz R, Pribaz JJ. Vascular considerations in composite midfacial allotransplantation. Plast Reconstr Surg. 2010 Feb;125(2):517-522. doi: 10.1097/PRS.0b013e3181c82e6f. PMID 19910848
- [Background] Rebergen SA, van der Wall EE, Doornbos J, de Roos A. Magnetic resonance measurement of velocity and flow: technique, validation, and cardiovascular applications. Am Heart J. 1993 Dec;126(6):1439-56. doi: 10.1016/0002-8703(93)90544-j. PMID 8249802
- [Background] Saliou G, Baledent O, Lehmann P, Paradot G, Gondry-Jouet C, Bouzerar R, Devisme G, Theaudin M, Deramond H, Le Gars D, Meyer ME, Vallee JN. [Acute CSF changes in the mesencephalon aqueduct after subarachnoid hemorrhage as measured by PC-MRI]. J Neuroradiol. 2009 Mar;36(1):41-7. doi: 10.1016/j.neurad.2008.07.004. Epub 2008 Aug 12. French. PMID 18701163
- [Background] Testelin, Sylvie, 2000. Incidence du flux microvasculaire sur le comportement des tissus transplantés. Exploration par vélocimétrie doppler laser. Université de Picardie Jules Verne-Amiens.
- [Background] Yim PJ, Tilara A, Nosher JL. The paradoxical flow hypothesis of the carotid artery: supporting evidence from phase-contrast magnetic resonance imaging. J Stroke Cerebrovasc Dis. 2008 Mar-Apr;17(2):101-8. doi: 10.1016/j.jstrokecerebrovasdis.2007.10.004. PMID 18346653
- [Background] Yzet T, Bouzerar R, Baledent O, Renard C, Lumbala DM, Nguyen-Khac E, Regimbeau JM, Deramond H, Meyer ME. Dynamic measurements of total hepatic blood flow with Phase Contrast MRI. Eur J Radiol. 2010 Jan;73(1):119-24. doi: 10.1016/j.ejrad.2008.09.032. Epub 2008 Nov 12. PMID 19008062